CLINICAL TRIAL: NCT04071899
Title: French Validation of a Severity Scale in REM Sleep Behavior Disorder
Brief Title: French Validation of a Severity Scale in REM Sleep Behavior Disorder (SEV-TCSP)
Acronym: SEV-TCSP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Société Française de Recherche et Médecine du Sommeil (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNI 2018 FANTINI (SEV-TCSP); 2018-A02473-52 (Other: ANSM)
Record Dates: First submitted 2019-07-29; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: REM Sleep Behavior Disorder
Keywords: REM Sleep Behavior Disorder; Validation scale
MeSH Terms: conditions — REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: patients with RBD
  Interventions: Other: Scale vaidation
- Bedpartners: Subjects which are the bedpartners of patients with RBD
  Interventions: Other: Scale vaidation

INTERVENTIONS:
Other: Scale vaidation — It's just filling a scale in order to validate it in French

SUMMARY:
REM (Rapid Eye Movements) Sleep Behavior Disorder (RBD) is a parasomnia characterized by episodes of elaborate or violent motor activity during dreams, which can lead to injury and sleep disruption in patient and / or his/her spouse. This is due to the loss of the normal muscle atonia during REM Sleep. RBD is often associated to neurodegenerative diseases, and may even precede them for several years as an early marker. Currently, there is no scale or tool for assessing the severity of RBD. Nevertheless, it is crucial to have a tool of severity when one wants to study the natural evolution of this disorder, as well as the possible effect of a drug in the context of a clinical trial. A Severity Scale of RBD has recently been proposed within the International RBD Study Group and an international validation study in several languages is being considered.

The main objective of this study is to validate a new scale of severity of the REM sleep behavior disorder (RBD Severity Scale or RBDSS) and to characterize its metrological properties, in particular its concurrent validity, internal consistency and reproducibility

DETAILED DESCRIPTION:
Research involving the human person, non-interventional, category 3

80 patients with RBD of any etiology (eg Idiopathic RBD, RBD associated with Parkinson's Disease, Multiple System Atrophy, Narcolepsy etc.) and their bedpartners (if available) will be include in 5 French centers (Clermont-Ferrand, Paris, Nantes, Montpellier et Lyon) Patients, and their bedpartners (if available), will be seen 2 times at 1 week intervals.

For the patients Visit 1 (Day 0): duration : 60 minutes

* Information to patient and collection of non-opposition
* Collection of socio-demographic data: age, sex, level of education
* Clinical data collection: duration of RBD, duration and severity of the concomitant disease:, medical and surgical history
* Assessment of cognitive functions: Mini Mental State Examination
* Verification of inclusion / exclusion criteria
* Ongoing treatments and calculation of Levodopa Equivalent Daily Dose (LEDD) for PD patients.
* RBD severity scale for Patient (RBDSS-PT) + Global Clinical Impression-Severity Scale

Visit 2 (J7) : duration : 20 minutes

* Ongoing treatments
* RBDSS PT + Global Clinical Impression-Severity Scale (CGI-S-PT)
* Patient will be given a Weekly Severity Agenda for 4 weeks plus a copy of the RBSSS-PT + Global Clinical Impression-Severity Scale

At home, patients will fill :

D8 à D36 :

• Weekly Severity Agenda (wRBDQ) for 4 weeks

D36 :

* RBDSS-PT + Clinical Global Impression-Severity These documents will be mailed back in a pre-payed envelop. For the Bed Partners Visit 1 (D0- baseline): duration: 30 minutes
* Information of and collection of non opposition
* Collection of socio-demographic data: age, sex, level of education
* Assessment of cognitive functions: Mini Mental State Examination
* Verification of inclusion / exclusion criteria
* Ongoing Treatments
* RBD severity scale of the bed partner (RBDSS BP)+ Global Clinical Impression-Severity Scale

Visit 2 (D7- retest) : duration : 20 minutes

* Ongoing treatments
* RBDSS-BP + Clinical Overall Impression Severity Scale
* Patient will be given a Weekly Joint Severity Agenda to be completed together with the patient, (wRBDQ) for 4 weeks, plus a copy of the RBDSS-BP + CGI-S-BP

At home: bedpartners will fill:

D8 à D36 :

• Weekly Severity Agenda for 4 weeks, in common with patient

D36 :

• RBDSS-BP + Impression Global Clinique-Severity scale These documents will be mailed back in a pre-payed envelop.

ELIGIBILITY:
Inclusion Criteria:

* RBD patients:

  * Men or women aged 30 to 80
  * Patients with idiopathic and secondary RBD (including RBD associated with Parkinson's disease, Narcolepsy, Multiple System Atrophy or other neurological diseases) diagnosed according to the latest international criteria Classification of Sleep Disorders (ICSD-3 ).
  * Cooperation and understanding to strictly comply with the conditions laid down in the protocol
  * Affiliated to a social security system
  * bedpartners
  * Men or women aged 30 to 80
  * Subjects sharing the same bed as the patient for ≥70% of the time (e.g. at least 5 nights / week, or 20 nights / month)
  * -Cooperation and understanding to strictly comply with the conditions described in the protocol
  * Affiliated to a social security system

Exclusion Criteria:

-- RBD patients:

* Clinically defined dementia according to the criteria of DSM-V2 (Major Neurocognitive Disorder)
* Untreated Obstructive Sleep Apnea Syndrome (OSAS) (with IAH> 15 / h at vPSG)
* Patients under tutorship or curatorship or safeguard of justice
* No change in treatment should have occurred during the 4 weeks prior to inclusion in the study and no change in treatment should be expected a priori within one week of inclusion
* Bedpartners
* Clinically defined dementia according to the criteria of DSM-V2 (Major Neurocognitive Disorder)
* Patients under tutorship or curatorship or safeguard of justice

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with RBD and their bedpartner
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-06-24 (Estimated); Study Completion 2020-09-24 (Estimated)

PRIMARY OUTCOMES:
French validation of a new scale of severity of REM Sleep behavior disorder for patient | Day 7
  The scale contains 8 items in the patient version. Each of them focusing on one RBD symptom, are evaluated in terms of their frequency and severity. This scale was administered at Day7 to evaluate concurrent validity, internal consistency and reproducibility
French validation of a new scale of severity of REM Sleep behavior disorder for patient | Day 0
  The scale contains 8 items in the patient version. Each of them focusing on one RBD symptom, are evaluated in terms of their frequency and severity. This scale was administered at Day 0 to evaluate concurrent validity, internal consistency and reproducibility

SECONDARY OUTCOMES:
French validation of a new scale of severity of REM Sleep behavior disorder for bedpartners | Day 7
  The scale contains 6 items in the patient version. After two introductory questions that are not scored, the scale includes items concerning the spouse's RBD symptoms and are evaluated in terms of their frequency and severity. This scale was administered at Day 7 to to evaluate concurrent validity, internal consistency and reproducibility
French validation of a new scale of severity of REM Sleep behavior disorder for bedpartners | Day 0
  The scale contains 6 items in the patient version. After two introductory questions that are not scored, the scale includes items concerning the spouse's RBD symptoms and are evaluated in terms of their frequency and severity. This scale was administered at Day 0 to to evaluate concurrent validity, internal consistency and reproducibility
Evaluation of the psychometric properties of the patient scale according to the etiology of the RBD | Day 7
  The total pool of patients will be divided into different groups according to the etiology (RBD-Idiopathic, RBD-parkinsons disease, RBD- Multiple System Atrophy, RBD-Narcolepsy etc.) and the validity in each condition will be evaluated
Evaluation of the fluctuations in the frequency and severity of RBD symptoms and their "night-to-night" variability through the collection of daily data over a four-week period | Day 28
  In order to control variability of symptoms, patients and their bed partners will complete a Weekly Symptom Diary (weekly-RBD Questionnaire), measuring the frequency and severity of symptoms daily for 4 weeks to determine the fluctuation of symptoms over a long period
Evaluation of the RBD severity using Clinical Global Impression-Severity | Day 7
  This scale is s the only currently available measure of severity of RBD. It includes 7 categories that are from 1 to 7: Normal (no symptoms), Minimal, Light, Moderate, Marked, Severe, Very Severe

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Livia Fantini, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (5):
- France (5):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital de la Croix Rousse, Lyon
  - Clinique beausoleil, Montpellier
  - CHU Nantes, Nantes
  - AP-HP, Paris

REFERENCES:
- [Derived] Fantini ML, Postuma RB, Puligheddu M, Rieu I, Venel E, Figorilli M, Cochen-DeCock V, Leclair-Visonneau L, Arnaldi D, Mattioli P, Peter-Derex L, Ricordeau F, Terzaghi M, Arnulf I, Stefani A, Videnovic A, Chirol C, Pereira B; International RBD Study Group. Validation of the International REM Sleep Behavior Disorder Study Group Symptoms Severity Scale (IRBD-SSS): a new tool to assess RBD clinical severity. J Neurol. 2024 Nov;271(11):7264-7271. doi: 10.1007/s00415-024-12702-9. Epub 2024 Sep 27. PMID 39327269